CLINICAL TRIAL: NCT00908908
Title: An Open-Label, Non-Randomized, Single-Center Study to Determine the Metabolism and Elimination of Carbon-14 Labeled Eribulin Acetate (14C-Eribulin) in Patients With Advanced Solid Tumors
Brief Title: A Study to Determine the Metabolism and Elimination of Carbon-14 Labeled Eribulin Acetate (14C-Eribulin) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-E044-103
Record Dates: First submitted 2009-05-20; First posted 2009-05-27 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Failure of Multiple Prior Chemotherapy Regimens
MeSH Terms: interventions — eribulin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: eribulin

INTERVENTIONS:
Drug: eribulin — Cycle 1 day 1: radio-labeled dose of 2 mg radioactive eribulin, followed by 1.4 mg/m^2 of non-radio-labeled eribulin thereafter on days 1 and 8 every 21 days.
  Other Names: E7389

SUMMARY:
The purpose of this study is to determine the metabolism and elimination of carbon-14 labeled eribulin acetate (14C-eribulin) in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study will be conducted in two phases, the initial Study phase to administer the radio-labeled 14C-eribulin and collection of PK samples, and the Extension Phase when the patients will continue to receive non-radio-labeled eribulin. In the initial Study phase, patients will receive a single 2 mg flat dose of 14C-eribulin (approximately 80 to 90 microCuries) administered on Cycle 1 Day 1 as an intravenous (IV) bolus injection or infusion over 2-5 minutes. Following this initial dose, patients will remain in the research unit until Day 8 to complete sample collections of urine, blood and feces for PK analysis and determination of 14C-eribulin concentrations between Days 1 and 8.

On Day 8 patients will be re-assessed and discharged, and return on day 15 for physical exam, adverse event evaluation, and lab tests. The patients will then enter the Extension Phase of the study and continue to receive on-radio-labeled eribulin at a dose of 1.4 mg/m^2 on Days 1 and 8 of every 21 day cycle.

ELIGIBILITY:
Inclusion criteria:

1. Patients must have a histologically or cytologically confirmed advanced solid tumor that has progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy). Patients with measurable tumors according to RECIST are desirable but not essential.
2. Patients must be aged 18 years or older.
3. Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0,1, or 2.
4. Patients must have adequate renal function as evidenced by serum creatinine ≤135 µM/L (≤1.5 mg/dL) or creatinine clearance >= 40 mL/minute (min).
5. Patients must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) >= 1.5 x 10^9/L and platelet count >= 100 x 10^9/L.
6. Patients must have adequate hepatic function as evidenced by bilirubin ≤ 1.5 times the upper limit of normal (ULN) and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3 x ULN (in the case of liver metastases ≤ 5 x ULN), unless there are bone metastases, in which case liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase.
7. Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or below, except for stable sensory neuropathy ≤ Grade 2 and alopecia.
8. Patients must be willing and able to comply with the study protocol for the duration of the study.
9. Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

1. Patients who have received any of the following treatments within the specified period before treatment start:

   * chemotherapy, radiation, or biological therapy within three weeks
   * hormonal therapy within one week
   * any investigational drug within 4 weeks
   * systemic unconventional or alternative therapies including, but not limited to, herbal remedies within 4 weeks
2. Have had radiation therapy encompassing > 30% of marrow.
3. Have received prior treatment with mitomycin C or nitrosourea.
4. Have had major surgery within 4 weeks before starting study treatment
5. Patients with pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
6. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (e.g., radiologic) and/or symptoms of brain metastases must be stable for at least 4 weeks.
7. Patients with meningeal carcinomatosis.
8. Patients who are receiving anti-coagulant therapy with warfarin or related compounds, other than for line patency, and cannot be changed to heparin-based therapy, are not eligible. If a patient is to continue on mini-dose warfarin, then the prothrombin time (PT) or international normalized ratio (INR) must be closely monitored.
9. Women who are pregnant or breast-feeding; women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test; women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Peri-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
10. Patients with severe/uncontrolled intercurrent illness/infection.
11. Significant cardiovascular impairment (history of congestive heart failure > New York Heart Association (NYHA) grade II, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia).
12. Patients with organ allografts requiring immunosuppression.
13. Patients with known positive HIV status.
14. Patients with pre-existing neuropathy > Grade 2.
15. Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative.
16. Patients who participated in a prior eribulin clinical trial, whether or not they received eribulin (E7389).
17. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Koetz, MSc, Study Director — Eisai Limited
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 1 center in The Netherlands during the period of Mar 2009 to Jun 2009.
Period: Overall Study
Arm/Group | Eribulin
Started | 6
Adverse Event | 0
Withdrawl by Subject | 0
Administrative/Other | 0
Physician Decision | 0
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eribulin
Number analyzed (Participants) | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Excretion Balance of Radio-labeled 14C-eribulin: Total Recovery of Radioactive Dose in Urine and Feces.
Time Frame: 312 hours postdose
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: percent recovery
Groups:
- 14C-eribulin/Eribulin: Cycle 1 Day 1: radio-labeled dose of 2 mg radioactive eribulin, followed by 1.4 mg/m^2 of non-radio-labeled eribulin thereafter on Days 1 and 8 every 21 days.
Arm/Group | 14C-eribulin/Eribulin
Number analyzed (Participants) | 6
percent recovery | 90.4 (11.73)

2. Primary Outcome: Pharmacokinetics: AUC (0-t) for Total Radioactivity in Plasma
Description: Area under the plasma concentration-time curve from time zero to last quantifiable plasma concentration measuring total radioactivity exposure.
Time Frame: Between Days 1 and 8 of Cycle 1
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: ng eq*hr/mL/mg
Arm/Group | 14C-eribulin/Eribulin
Number analyzed (Participants) | 6
ng eq*hr/mL/mg | 269 (153.4)

3. Primary Outcome: Pharmacokinetics AUC (0-t) for Eribulin in Plasma
Description: Area under the plasma concentration-time curve from time zero to last quantifiable plasma concentration measuring exposure to eribulin.
Time Frame: Between Days 1 and 8 of Cycle 1
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: ng eq*hr/mL/mg
Arm/Group | 14C-eribulin/Eribulin
Number analyzed (Participants) | 6
ng eq*hr/mL/mg | 301 (164.9)

ADVERSE EVENTS:
Arm/Group | Eribulin
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin (N=6)
Headache (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1
Scab (Skin and subcutaneous tissue disorders) | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No